CLINICAL TRIAL: NCT02515357
Title: The MIMOSA (Mediterranean Diet/Lifestyle Intervention for the Management of Obstructive Sleep Apnea) Study
Brief Title: Mediterranean Diet/Lifestyle Intervention in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Meropi Kontogianni, Assistant Professor of Clinical Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Disorders; Metabolic Syndrome; Mediterranean Diet; Mediterranean Lifestyle
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders; Metabolic Syndrome | interventions — Standard of Care; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Placebo Comparator): This arm will receive standard care, i.e. CPAP prescription and brief written healthy lifestyle advice.
  Interventions: Behavioral: Standard care
- Mediterranean lifestyle group (Experimental): This arm will receive a hypocaloric diet and attend a comprehensive 6-month lifestyle intervention based on the Mediterranean lifestyle on top of standard care.
  Interventions: Behavioral: Mediterranean lifestyle
- Mediterranean diet group (Experimental): This arm will receive a hypocaloric diet and attend a comprehensive 6-month dietary intervention based on the Mediterranean dietary pattern on top of standard care.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Mediterranean lifestyle — Comprehensive 6-month lifestyle intervention (7 60-min group counselling sessions) aiming at promoting adherence to the Mediterranean lifestyle (food and food group consumption according to the Mediterranean diet, beneficial culinary practices, seasonality and locality of foods consumed, socialization during meals, adequate rest during the day through night sleep and siesta nap, sleep hygiene recommendations and adoption of a physically active lifestyle) and at achieving a 5-10% weight loss.
  Arms: Mediterranean lifestyle group
Behavioral: Standard care — General written instructions regarding the adoption of a healthy lifestyle.
  Arms: Control group
Behavioral: Mediterranean diet — Comprehensive 6-month lifestyle intervention (7 60-min group counselling sessions) aiming at promoting adherence to the Mediterranean dietary pattern (food and food group consumption according to the Mediterranean diet, beneficial culinary practices and seasonality and locality of foods consumed) and at achieving a 5-10% weight loss.
  Arms: Mediterranean diet group

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder characterized by recurrent episodes of partial or complete collapse of the upper airway during sleep, leading to pauses of breathing and arousals. Although previously considered as a local abnormality of the respiratory track, it is nowadays recognized as a systemic disease and an important cause of morbidity and mortality, since it is strongly associated with obesity (especially abdominal obesity) and cardiometabolic diseases, including cardiovascular diseases and diabetes mellitus. Interestingly, recent hypotheses support that the metabolic syndrome pathology, including insulin resistance, inflammation and oxidative stress may be involved in OSA pathogenesis. The modification of lifestyle habits, e.g. in terms of diet and physical activity, is currently explored as a mean of managing the disease in combination with the first line treatment, i.e., the application of continuous positive airway pressure (CPAP) during sleep. The available data support that weight loss, achieved through lifestyle modification, effectively reduces the severity of OSA and improves the associated cardiometabolic disorders in overweight or obese patients. However, studies exploring the potential effect of diet's quality or other lifestyle habits (such as physical activity) on OSA severity, besides weight loss, are currently lacking. Given that a Mediterranean dietary pattern, as well as other lifestyle habits adopted by the populations in the Mediterranean region, have been proven beneficial both for the prevention and the resolution of the metabolic syndrome and its associated cardiometabolic diseases, the aim of the present randomized, controlled, single-blind study is to implement an intensive intervention based on the Mediterranean lifestyle (hypocaloric diet and 7 group lifestyle counselling sessions) and to evaluate its potential benefits, compared with standard care (hypocaloric diet and written advice for healthy lifestyle), in a sample of patients with OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a chronic disease characterized by recurrent complete or partial interruptions of breathing during sleep due to obstruction of the upper airways, which leads to disturbances in gas exchange, hypoxia and consequent arousals. Beyond its adverse impact on sleep duration, sleep quality, as well as the functionality and cognitive function during the day (typical symptoms include fatigue, sleepiness, decreased reflexes, impaired memory, etc.). OSA is currently recognized as a major cause of morbidity and mortality due to its strong association with obesity and cardiometabolic diseases, including the metabolic syndrome (and its individual components, namely abdominal adiposity, impaired fasting glucose, dyslipidaemia and hypertension), cardiovascular diseases and diabetes mellitus. According to epidemiological data, its prevalence ranges from 2% to 7% in the general population (with a clear lead of obese middle-aged men), however it is estimated that a large proportion of patients (70-80%) remain undiagnosed making the disease a major public health challenge for the 21st century. Currently, the first line treatment for the management of moderate-to-severe OSA or mild OSA accompanied by symptoms (such as daytime sleepiness and cognitive disorders) and other diseases (such as hypertension and heart disease) is the application of continuous positive airway pressure (CPAP) during sleep, usually via a renal mask. CPAP has been proven effective in alleviating the symptoms of the disease (e.g. pauses of breathing during sleep and daytime sleepiness), however it is also characterized by high rates of non-compliance and its effectiveness in improving cardiometabolic indices has not yet been confirmed.

Given the strong relationship of OSA with obesity and its concomitant metabolic disorders, as well as the aforementioned restrictions of the use of CPAP as the sole treatment for the disease, lifestyle changes have currently emerged as a promising treatment for OSA. Indeed, several interventional studies have investigated the effect of lifestyle changes on the treatment of OSA, focusing primarily on weight loss - achieved through a hypocaloric diet, either solely or in combination with exercise and lifestyle counselling - and the available data support its effectiveness in reducing the severity of the disease and improving its associated cardiometabolic disorders in overweight patients. However, studies exploring the potential effect of diet's quality or other lifestyle habits (such as physical activity) on OSA severity and associated disorders, besides weight loss, are currently lacking. Given that a Mediterranean dietary pattern, as well as other lifestyle habits adopted by the populations in the Mediterranean region, have been proven beneficial both for the prevention and the resolution of the metabolic syndrome and its associated cardiometabolic diseases, the aim of the present study is to implement an intervention based on the Mediterranean lifestyle and to evaluate its potential beneficial effect on biochemical and clinical characteristics of a sample of patients with OSA, compared with standard care. In addition, the superiority of a lifestyle intervention based on the Mediterranean lifestyle to a dietary intervention based only on the Mediterranean diet will be explored, in order to evaluate possible beyond-diet benefits of the health-promoting lifestyle of the Mediterranean that also included reguiar physical activity, adequate rest during the day, conviviality, etc.

This study will be a randomized, controlled, single-blind clinical trial. The study sample will consist of adult (18-65 year old), overweight or obese (Body Mass Index > 25 kg/m2) patients with moderate or severe OSA (Apnea Hypopnea Index > 15 events/hour) confirmed through polysomnography at the Center of Sleep Disorders of the 1st Department of Critical Care and Pulmonary Services of "Evaggelismos" General Hospital of Athens. At baseline, patients will be informed in detail about the study and will give their written consent. Then, subjects will be randomly assigned to one of 3 groups: (a) the control group, receiving CPAP therapy and written general advice for a healthy lifestyle, (b) the Mediterranean diet group (MDG), participating in a 6-month comprehensive weight-loss dietary intervention based on the Mediterranean dietary pattern, and (c) the Mediterranean lifestyle group (MLG), receiving the same intensive dietary intervention as the MDG in addition to other healthy behaviours incorporated in the traditional lifestyle of the Mediterranean.

Patients allocated in the two intensive intervention arms will attend a comprehensive intervention, comprising seven 60-min group counselling sessions (up to 5 patients per group) carried out in the laboratory of Clinical Nutrition & Dietetics of Harokopio University of Athens under the supervision of experienced clinical dietitians, conducted every two weeks for the first 2 months and every month for the following 4 months until the end of the 6-month intervention. For both the MDG and the MLG, the intervention will aim at a 5-10% weight loss during the 6-month period and an increase in the level of adherence to the plant-based Mediterranean diet. Specifically, all food groups of the Mediterranean diet will be targeted according to the pattern proposed in the Mediterranean diet pyramid (e.g. increase in the consumption of fruits, vegetables, whole grains and legumes, decrease in the consumption of red meat and sweets, preference in olive oil as the main source of dietary fat, prudent alcohol consumption, etc.), while beneficial culinary practices, as well as seasonality and locality of food products consumed, will also be addressed. Patients allocated in the MLG will additionally receive counselling on other lifestyle habits, with emphasis on adopting a physically active lifestyle and achieving adequate rest during the day (both night sleep and siesta nap), as parts of the healthy Mediterranean lifestyle. Dietary or lifestyle counselling will be based on the goal setting theory, while motivational and behavioural strategies will also be used.

The assessment of patients' clinical, laboratory and lifestyle characteristics will be performed at baseline, at the end of the 6-month intervention and 1 year after the study entry at the Center of Sleep Disorders of the 1st Department of Critical Care and Pulmonary Services of "Evaggelismos" General Hospital of Athens. The evaluation will include: 1) brief medical history assessment, 2) assessment of the severity of the disease through polysomnography, 3) evaluation of insomnia through the Athens Insomnia Scale, 4) assessment of daytime sleepiness through the Epworth Sleepiness Scale, 5) evaluation of the quality of life through the SF-36 questionnaire, 6) dietary assessment through a semiquantitative food frequency questionnaire (data from the food frequency questionnaire will be used to evaluate participants' food group and individual food and beverage consumption, as well as their adherence to the Mediterranean diet through the Mediterranean Diet Score) and 24-hour dietary recalls (data from the 24-h dietary recalls will be analysed in terms of energy, macro- and micronutrient intake using the Nutritionist Pro, version 2.2 software, as well as of meal frequency and patterns), 7) physical activity assessment through the International Physical Activity Questionnaire, 8) anthropometric measurements (height, weight, waist and hip circumference), 9) blood pressure measurement and 10) fasting blood sample and urine sample collection for laboratory measurements (lipid profile, markers of glucose metabolism, markers of liver function, inflammatory markers, markers of oxidative stress, etc.) using automated analysers and/or commercial ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of obstructive sleep apnea diagnosed through polysomnography
2. Presence of overweight or obesity (Body Mass Index > 25 kg/m2)

Exclusion Criteria:

1. Presence of central sleep apnea
2. Presence of other causes of sleep disorders, such as narcolepsy, restless leg syndrome or chronic pain syndrome
3. Hospitalization during the last year due to acute or chronic respiratory disease or required use of supplemental oxygen
4. Presence of diabetes mellitus
5. Presence of cardiovascular disease
6. Presence of severe hypertension (blood pressure > 160/95 mm Hg)
7. Presence of neoplasm
8. Presence of chronic inflammatory diseases
9. Presence of psychiatric disorders, such as major depression, schizophrenia or suicidal ideation
10. Pregnancy or breast feeding (for women)
11. Surgery during the last three months
12. Reception of antipsychotics, antidepressants or other sleep inducing drugs, systematic reception of steroids or hormone replacement therapy for women
13. Excessive alcohol consumption (> 210 or > 140 gr of alcohol per week for men and women, respectively)
14. Adherence to a hypocaloric diet for weight loss or changes in dietary habits during the last six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Severity of obstructive sleep apnea | 6 months
  Reduction in the Apnea Hypopnea Index (AHI)

SECONDARY OUTCOMES:
Sleep quality | 6 months
  Improvement in the Athens Insomnia Scale score
Daytime sleepiness | 6 months
  Reduction in the Epworth Sleepiness Scale score
Physical and mental health | 6 months
  Improvement in physical and mental health scales assessed through the SF-36 questionnaire
Insulin resistance | 6 months
  Reduction in Homeostasis Model of Assessment of Insulin Resistance (HOMA-IR)
Subclinical inflammation | 6 months
  Reduction in circulation c-reactive protein (CRP) and tumour necrosis factor a (TNF-a) levels, and increase in circulating adiponectin levels
Oxidative stress | 6 months
  Reduction in urine 8-isoprostane and 8OHd-guanosine levels
Metabolic syndrome prevalence (%) | 6 months
  Reduction in the prevalence of the metabolic syndrome defined according to the criteria proposed by Alberti et al. 2009 (presence of at least three of the following: increased waist circumference, increased triglycerides, decreased high-density lipoprotein cholesterol, hyperglycemia and hypertension)

CONTACTS AND LOCATIONS:
Overall Officials: Meropi D Kontogianni, PhD, Study Director — Harokopio University
Locations (1):
- Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Data will be available upon demand.

REFERENCES:
- [Derived] Georgoulis M, Yiannakouris N, Kechribari I, Lamprou K, Perraki E, Vagiakis E, Kontogianni MD. Sustained improvements in the cardiometabolic profile of patients with obstructive sleep apnea after a weight-loss Mediterranean diet/lifestyle intervention: 12-month follow-up (6 months post-intervention) of the "MIMOSA" randomized clinical trial. Nutr Metab Cardiovasc Dis. 2023 May;33(5):1019-1028. doi: 10.1016/j.numecd.2023.02.010. Epub 2023 Feb 18. PMID 36958969
- [Derived] Georgoulis M, Yiannakouris N, Kechribari I, Lamprou K, Perraki E, Vagiakis E, Kontogianni MD. Dose-response relationship between weight loss and improvements in obstructive sleep apnea severity after a diet/lifestyle interventions: secondary analyses of the "MIMOSA" randomized clinical trial. J Clin Sleep Med. 2022 May 1;18(5):1251-1261. doi: 10.5664/jcsm.9834. PMID 34915980
- [Derived] Georgoulis M, Yiannakouris N, Tenta R, Fragopoulou E, Kechribari I, Lamprou K, Perraki E, Vagiakis E, Kontogianni MD. A weight-loss Mediterranean diet/lifestyle intervention ameliorates inflammation and oxidative stress in patients with obstructive sleep apnea: results of the "MIMOSA" randomized clinical trial. Eur J Nutr. 2021 Oct;60(7):3799-3810. doi: 10.1007/s00394-021-02552-w. Epub 2021 Apr 10. PMID 33839919
- [Derived] Georgoulis M, Yiannakouris N, Kechribari I, Lamprou K, Perraki E, Vagiakis E, Kontogianni MD. The effectiveness of a weight-loss Mediterranean diet/lifestyle intervention in the management of obstructive sleep apnea: Results of the "MIMOSA" randomized clinical trial. Clin Nutr. 2021 Mar;40(3):850-859. doi: 10.1016/j.clnu.2020.08.037. Epub 2020 Sep 6. PMID 32928580